CLINICAL TRIAL: NCT03627585
Title: Reprogramming to Prevent Progressive Pacemaker-Induced Remodelling
Acronym: PPPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, KK Witte, Senior Lecturer in Cardiology, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICA-CDRF-2016-02-055
Record Dates: First submitted 2018-08-06; First posted 2018-08-13 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Left Ventricular Dysfunction; Heart Failure, Systolic; Left Ventricular Failure; Pacemaker; Complication, Mechanical
Keywords: pacemaker; heart failure; left ventricular dysfunction; bradycardia; remodelling
MeSH Terms: conditions — Ventricular Dysfunction, Left; Heart Failure, Systolic; Heart Failure; Bradycardia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Patients received echocardiogram but no pacemaker reprogramming or personalisation.
- Personalised programming (Active Comparator): Patient will have tailored pacemaker programming based on echocardiographic findings, blood results, and symptoms in an attempt to minimise right ventricular pacing and extend battery longevity.
  Interventions: Device: Personalised programming

INTERVENTIONS:
Device: Personalised programming — Reprogramming protocol already test in an observation cohort will be utilised which will direct physiologists to consider pacemaker mode, base rate, utilisation of rate response, hysteresis, sleep and rest rates as well as lead outputs.
  Arms: Personalised programming

SUMMARY:
The aim is to provide evidence of the long-term benefits of personalised pacemaker programming on heart function and battery longevity.

This will be achieved by showing in a single centre, phase II, double-blind, randomised, placebo-controlled trial that reducing the amount of pacemaker beats to a minimum reverses these changes and extends battery life.

DETAILED DESCRIPTION:
Patients (n=70) with long-term (>2 years) permanent pacemakers with avoidable RV pacing will be invited to participate in a single-centre, phase II, randomised, double-blind placebo-controlled trial of optimised pacing programming versus standard care. Those randomised to the intervention arm will have personalised programming to avoid right ventricular pacing, whilst those allocated to standard care will have no programming changes made. All participants will be invited back at 6 months for a repeat echocardiogram, quality of life assessment (EQ-5D-5L), blood tests and pacemaker check.

ELIGIBILITY:
Inclusion Criteria:

* Chronic right ventricular bradycardia pacemaker implanted for at least 24 months
* Willing and able to give informed consent for the intervention

Exclusion Criteria:

* Known poor imaging quality patients (details of patients excluded for this reason will be recorded)
* Patients with complete heart block and no reprogramming options

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-01-06 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | 6 months
  Left ventricular functional measure using either 3D volumes or Simpson's Biplane obtained from echocardiographic images.

SECONDARY OUTCOMES:
LV remodelling parameters | 6 months
  left ventricular end diastolic and systolic volumes
Quality of Life Measures | 6 months
  EQ-5D, Minnesota living with Heart Failure Questionnaire
Battery Longevity | 6 months
  Impedance

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Witte, MD, Principal Investigator — University of Leeds
Locations (2):
- United Kingdom (2):
  - Harrogate District Foundation Trust, Harrogate
  - Leeds Teaching Hospitals NHS Trust, Leeds

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Paton MF, Gierula J, Lowry JE, Cairns DA, Bose Rosling K, Cole CA, McGinlay M, Straw S, Byrom R, Cubbon RM, Kearney MT, Witte KK. Personalised reprogramming to prevent progressive pacemaker-related left ventricular dysfunction: A phase II randomised, controlled clinical trial. PLoS One. 2021 Dec 13;16(12):e0259450. doi: 10.1371/journal.pone.0259450. eCollection 2021. PMID 34898655